CLINICAL TRIAL: NCT06197022
Title: Scoring-Balloon Angioplasty and Sirolimus-Eluting Balloon Angioplasty for the Treatment of Diffuse, Small Vessel Coronary Artery Disease (SCA-DEB Study)
Acronym: SCA-DEB
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University National Heart Hospital (Other)
Collaborators: Meril Life Sciences Pvt. Ltd. (Industry)
Responsible Party: Principal Investigator, Dobrin Vassilev, Professor, Medica Cor Heart Hospital
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCA-DEB_2022
Record Dates: First submitted 2023-12-25; First posted 2024-01-09 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2023-12

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Scoring Balloon Angioplasty (Other): Combination of scoring-balloon angioplasty (SBA) plus sirolimus-eluting balloon angioplasty (SEBA) for diffuse (lesion length ≥20 mm), small vessel (diameter 1.5 mm -2.75 mm) coronary disease.
  Interventions: Device: Mozec™ SEB Sirolimus Eluting Rx PTCA Balloon Dilatation Catheter

INTERVENTIONS:
Device: Mozec™ SEB Sirolimus Eluting Rx PTCA Balloon Dilatation Catheter — Combination of scoring-balloon angioplasty (SBA) plus sirolimus-eluting balloon angioplasty (SEBA) for diffuse (lesion length ≥20 mm), small vessel (diameter 1.5 mm -2.75 mm) coronary disease.

SUMMARY:
This is a prospective, single-center, single-arm study to evaluate the feasibility and safety of the combination of Scoring-Balloon Angioplasty and Sirolimus-Eluting Balloon Angioplasty for the treatment of diffuse, small vessel coronary artery disease. The objective of the study is to demonstrate the feasibility and safety of the combination of scoring-balloon angioplasty (SBA) plus sirolimus-eluting balloon angioplasty (SEBA) for diffuse (lesion length ≥20 mm), small vessel (diameter 1.5 mm -2.75 mm) coronary disease.

ELIGIBILITY:
Inclusion Criteria:

1. Patientsaged≥18years.
2. Presence of epicardial coronary artery disease with lesion length ≥ 20 mm and vessel diameter less than 2.75 mm and more than 1.5 mm with diameter stenosis >50% by visual evaluation.

Exclusion Criteria:

1. Life expectancy < 2 years
2. Left ventricular EF ≤40%
3. Pregnantorlactatingfemales.
4. Moderate and moderate-to-severe valvular heart disease.
5. Hemodynamic instability.
6. Severe renal dysfunction, defined as an eGFR <30 mL/min/1.73 m2
7. Patients with hypersensitivity or allergies to aspirin, heparin, clopidogrel, ticlopidine, bivalirudin, prasugrel, ticagrelor and drug such as Sirolimus (Rapamycin) or similar drugs or any analogue or derivative, hydrogenated castor oil, PVP or any contrast media.
8. Patients in whom anti-platelet and/or anti-coagulant therapy are contraindicated.
9. Patients judged to have a lesion that prevents complete inflation of an angioplasty balloon.
10. Transplant patients.
11. Patients with calcified lesion requiring other type of treatment such as Rotational Atherectomy.
12. Unprotected left main coronary artery lesions
13. Coronary artery spasm in the absence of a significant stenosis.
14. Patients whose diseased segment cannot be pre-dilated or prepared before drug coated balloon treatment.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 106 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Major Adverse Cardiovascular Events (MACE) | 12 months
  Composite of non-fatal MI, cardiovascular death, and target lesion revascularization

SECONDARY OUTCOMES:
Cardiovascular Death | 3 months, 6 months, 12 months, 24 months, 36 months
  Defined as per Academic Research Consortium-2 (ARC-2) criteria
Non-fatal Myocardial Infarction | 3 months, 6 months, 12 months, 24 months, 36 months
  Non-fatal myocardial infarction (MI) is defined as per the fourth universal definition of MI
Target Lesion Revascularization (TLR) | 3 months, 6 months, 12 months, 24 months, 36 months
  It is defined as repeat percutaneous intervention of the target lesion or bypass surgery of the target vessel performed for restenosis or other complication of the target lesion
Target Vessel Failure (TVF) | 3 months, 6 months, 12 months, 24 months, 36 months
  It is defined as the composite of cardiovascular death, target vessel myocardial infarction and target vessel revascularization
Restenosis | 3 months
  Defined as >50% stenosis at the treated segment.
Major bleeding | 3 months, 6 months, 12 months, 2 years and 3 years
  Defined as bleeding that causes hemodynamic instability and/or leads to blood transfusion
Quality of Life Score | Baseline, 3 months, 6 months, 12 months
  OverallHealthStatusassessedbyShortFormSurvey(SF-12)
Device success | During the procedure
  Defined as the ability of the study device to be delivered, dilated, and retrieved from the target lesion

CONTACTS AND LOCATIONS:
Locations (1):
- Medica Core Heart Hopsital, Rousse, Bulgaria

IPD SHARING:
Plan to Share IPD: Undecided